CLINICAL TRIAL: NCT02018887
Title: A Single- and Multiple-Ascending Dose, Safety, Tolerability,Pharmacokinetic and Pharmacodynamic Study of LY2969822 in Healthy Subjects
Brief Title: A Study of LY2969822 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15259; I4W-FW-HMJD (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-12-12; First posted 2013-12-23 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY2969822 (Part A) (Experimental): Single dose of LY2969822 administered orally in 2 of 3 study periods.
  Interventions: Drug: LY2969822
- Placebo (Part A) (Placebo Comparator): Single dose of placebo administered orally in 1 of 3 study periods.
  Interventions: Drug: Placebo
- LY2969822 (Part B) (Experimental): LY2969822 administered orally for 14 days.
  Interventions: Drug: LY2969822
- Placebo (Part B) (Placebo Comparator): Placebo administered orally for 14 days.
  Interventions: Drug: Placebo
- LY2969822 (Part C) (Experimental): LY2969822 administered orally for 14 days.
  Interventions: Drug: LY2969822
- Placebo (Part C) (Placebo Comparator): Placebo administered orally for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2969822 — Capsules administered orally
  Arms: LY2969822 (Part A); LY2969822 (Part B); LY2969822 (Part C)
Drug: Placebo — Capsules administered orally
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C)

SUMMARY:
The purpose of this study is to evaluate how safe LY2969822 (study drug) is and whether it causes any side effects. The study will also measure how much of the study drug gets into the blood stream and how long it takes the body to get rid of the study drug. This is the first time that this study drug is being given to participants. This study is for research purposes only and is not intended to treat any medical condition.

DETAILED DESCRIPTION:
Participants in Part A will complete three study periods, which together will last about 40 days. Participants in Parts B and C will complete one study period which will last about 17 days, but the total study time is about 40 days. Each participant may only enroll in one part. Screening is required within 28 days prior to the start of the study for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Male participants must agree to use a reliable method of birth control in addition to having their partner use another method for the duration of the study and for 3 months after the last dose of LY2969822
* Female participants must not be of child-bearing potential
* Participants have a body mass index (BMI) of 18.5 to 29.9 kilogram per meter square (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Have participated, within the last 30 days (prior to first dose in this study), in a clinical trial involving an investigational product
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Intended use of over-the-counter medication within 14 days prior to dosing or during the study with the exception of vitamins and mineral supplements or occasional paracetamol or acetaminophen
* Intended use of herbal supplements or prescription medications, other than stable doses of thyroid or estrogen hormone replacement, within 14 days prior to dosing or during the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had 3 parts. Part A-Single ascending dose, 3-period, crossover study (Cohorts 1-2). Part B-Multiple ascending dose, parallel study (Cohorts 3-7). Part C-Multiple dose, single dose level study (Cohort 8). Each participant enrolled in 1 cohort. Replacement participants received interventions intended for those that discontinued early.
Groups:
- Part A: Cohort 1: Participants were randomised to receive 2 single, oral doses of LY2969822 and 1 oral dose of placebo over the 3 study periods in a crossover fashion. For each study period, it was intended that 6 subjects would receive LY2969822 and 3 subjects would receive placebo.
  Placebo administered once, orally (PO) at all three periods. 2 milligrams (mg) LY2969822 administered once, PO during period 1. 20 mg LY2969822 administered once, PO during period 2. 40 mg LY2969822 administered once, PO during period 3.
- Part A: Cohort 2: Participants were randomised to receive 2 single, oral doses of LY2969822 and 1 oral dose of placebo over the 3 study periods in a crossover fashion. For each study period, it was intended that 6 subjects would receive LY2969822 and 3 subjects would receive placebo.
  Placebo administered once, PO at all three periods. 6 mg LY2969822 administered once, PO during period 1. 60 mg LY2969822 administered once, PO during period 2. 20 mg LY2969822 administered once, PO during period 3.
- Cohorts 3-7 - Placebo: Placebo administered once a day (QD) or twice a day (BID), PO, for 14 days.
- Cohort 3 - 20 mg LY2969822 QD: 20 mg LY2969822 administered QD, PO, for 14 days.
- Cohort 4 - 40 mg LY2969822 QD Titrated: Up to 40 mg LY2969822 administered QD, PO, for 14 days. Titration: 6 mg QD for 3 days, 20 mg QD for 2 days, and 40 mg QD for 9 days.
- Cohort 5 - 80 mg LY2969822 QD Titrated: Up to 80 mg LY2969822 administered QD, PO, for 14 days. Titration: 6 mg QD for 2 days, 20 mg QD for 2 days, 40 mg QD for 2 days and 80 mg QD for 8 days.
- Cohort 6 - 80 mg LY2969822 BID Titrated: Up to 80 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, 40 mg BID for 2 days, and 80 mg BID for 6 days.
- Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated: Up to 40 mg LY2969822 administered BID, PO, for 14 days. Titration: 10 mg BID for 1 day, 20 mg BID for 1 day, and 40 mg BID for 12 days.
- Cohort 8 - Placebo BID: Placebo administered BID, PO, for 14 days.
- Cohort 8A - 40 mg LY2969822 BID Titrated: Up to 40 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, and 40 mg BID for 8 days.)
- Cohort 8B - 20 mg LY2969822 BID Titrated: Up to 20 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, and 20 mg BID for 10 days.
Period: Part A: Cohorts 1-2: Period 1
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Cohorts 3-7 - Placebo | Cohort 3 - 20 mg LY2969822 QD | Cohort 4 - 40 mg LY2969822 QD Titrated | Cohort 5 - 80 mg LY2969822 QD Titrated | Cohort 6 - 80 mg LY2969822 BID Titrated | Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated | Cohort 8 - Placebo BID | Cohort 8A - 40 mg LY2969822 BID Titrated | Cohort 8B - 20 mg LY2969822 BID Titrated
Started | 9 | 9 | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.)
Received One Dose of Study Drug | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohorts 1-2: Period 2
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Cohorts 3-7 - Placebo | Cohort 3 - 20 mg LY2969822 QD | Cohort 4 - 40 mg LY2969822 QD Titrated | Cohort 5 - 80 mg LY2969822 QD Titrated | Cohort 6 - 80 mg LY2969822 BID Titrated | Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated | Cohort 8 - Placebo BID | Cohort 8A - 40 mg LY2969822 BID Titrated | Cohort 8B - 20 mg LY2969822 BID Titrated
Started | 9 | 9 | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.)
Received One Dose of Study Drug | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohorts 1-2: Period 3
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Cohorts 3-7 - Placebo | Cohort 3 - 20 mg LY2969822 QD | Cohort 4 - 40 mg LY2969822 QD Titrated | Cohort 5 - 80 mg LY2969822 QD Titrated | Cohort 6 - 80 mg LY2969822 BID Titrated | Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated | Cohort 8 - Placebo BID | Cohort 8A - 40 mg LY2969822 BID Titrated | Cohort 8B - 20 mg LY2969822 BID Titrated
Started | 9 | 9 | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.)
Received One Dose of Study Drug | 8 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 8 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Cohorts 3-7 Overall
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Cohorts 3-7 - Placebo | Cohort 3 - 20 mg LY2969822 QD | Cohort 4 - 40 mg LY2969822 QD Titrated | Cohort 5 - 80 mg LY2969822 QD Titrated | Cohort 6 - 80 mg LY2969822 BID Titrated | Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated | Cohort 8 - Placebo BID | Cohort 8A - 40 mg LY2969822 BID Titrated | Cohort 8B - 20 mg LY2969822 BID Titrated
Started | 0 (Column for Part A data only.) | 0 (Column for Part A data only.) | 15 | 9 | 9 | 9 | 9 | 9 | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.)
Received at Least One Dose of Study Drug | 0 | 0 | 15 | 9 | 9 | 9 | 9 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 15 | 9 | 8 | 9 | 8 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0
Period: Part C: Cohort 8 Overall
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Cohorts 3-7 - Placebo | Cohort 3 - 20 mg LY2969822 QD | Cohort 4 - 40 mg LY2969822 QD Titrated | Cohort 5 - 80 mg LY2969822 QD Titrated | Cohort 6 - 80 mg LY2969822 BID Titrated | Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated | Cohort 8 - Placebo BID | Cohort 8A - 40 mg LY2969822 BID Titrated | Cohort 8B - 20 mg LY2969822 BID Titrated
Started | 0 | 0 | 0 (Placebo was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 0 (This dose was not administered in this period.) | 10 | 4 | 7
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 4 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A: Cohorts 1-2: Part A Single Ascending Dose (SAD): Cohort 1 received placebo, 2 mg, 20 mg, or 40 mg LY2969822 PO, once, in each of 3 study periods. Cohort 2 received placebo, 6 mg, 60 mg, or 20 mg LY2969822 PO, once, in each of 3 study periods. At least 5 days elapsed between doses of study drug.
- Part B: Placebo; Part B: Cohorts 3; Part B: Cohorts 4; Part B: Cohorts 5; Part B: Cohorts 6; Part B: Cohorts 7: Part B Multiple Ascending Dose (MAD): Participants were assigned to 1 of 5 dosing cohorts (Cohorts 3 - 7). Cohort 3 received either placebo or 20 mg LY2969822 QD, PO, for 14 days. Cohort 4 received either placebo or up to 40 mg LY2969822 QD, PO, for 14 days (Titration: 6 mg QD for 3 days; 20 mg QD for 2 days, and 40 mg QD for 9 days.) Cohort 5 received placebo or up to 80 mg LY2969822 QD, PO, for 14 days. (Titration: 6 mg QD for 2 days; 20 mg QD for 2 days; 40 mg QD for 2 days and 80 mg QD for 8 days.) Cohort 6 received either placebo or up to 80 mg LY2969822 BID, PO for 14 days. (Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, 40 mg BID for 2 days, and 80 mg BID for 6 days.) Cohort 7 received either placebo or up to 40 mg LY2969822 BID, PO for 14 days with rapid titration. (Titration: 10 mg BID for 1 day, 20 mg BID for 1 day, 40 mg BID for 12 days.)
- Part C: Cohort 8: Part C Multiple Dose, Single Dose Level: Cohort 8A received either placebo or up to 40 LY2969822 BID, PO, for 14 days. (Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, and 40 mg BID for 8 days.) Cohort 8B received either placebo or up to 20 mg LY2969822 BID, PO, for 14 days. (Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, and 20 mg BID for 10 days.)
- Total: Total of all reporting groups
Arm/Group | Part A: Cohorts 1-2 | Part B: Placebo | Part B: Cohorts 3 | Part B: Cohorts 4 | Part B: Cohorts 5 | Part B: Cohorts 6 | Part B: Cohorts 7 | Part C: Cohort 8 | Total
Number analyzed (Participants) | 18 | 15 | 9 | 9 | 9 | 9 | 9 | 21 | 99
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part A | 35.1 (9.5) | NA (NA) — Part A:Cohorts 1-2 data only. | NA (NA) — Part A:Cohorts 1-2 data only. | NA (NA) — Part A:Cohorts 1-2 data only. | NA (NA) — Part A:Cohorts 1-2 data only. | NA (NA) — Part A:Cohorts 1-2 data only. | NA (NA) — Part A:Cohorts 1-2 data only. | NA (NA) — Part A:Cohorts 1-2 data only. | 35.1 (9.5)
  Part B | NA (NA) — Part B: Cohorts 3-7 data only. | 32.6 (7.6) | 32.7 (7.4) | 34.6 (6.8) | 32.2 (6.7) | 31.6 (5.7) | 35.1 (10.6) | NA (NA) — Part B: Cohorts 3-7 data only. | 33.1 (7.4)
  Part C | NA (NA) — Part C: Cohort 8 data only. | NA (NA) — Part C: Cohort 8 data only. | NA (NA) — Part C: Cohort 8 data only. | NA (NA) — Part C: Cohort 8 data only. | NA (NA) — Part C: Cohort 8 data only. | NA (NA) — Part C: Cohort 8 data only. | NA (NA) — Part C: Cohort 8 data only. | 40.3 (5.3) | 40.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 18 | 15 | 9 | 9 | 9 | 9 | 9 | 21 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 15 | 9 | 9 | 9 | 9 | 9 | 21 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 14 | 9 | 8 | 9 | 8 | 9 | 21 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 18 | 15 | 9 | 9 | 9 | 9 | 9 | 21 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other nonserious adverse events (AEs) and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Through End of Study (up to Week 7)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 1 - Placebo; Cohort 2 - Placebo: Placebo administered once, PO.
- Cohort 1 - 2 mg LY2969822; Cohort 1 - 20 mg LY2969822; Cohort 2 - 20 mg LY2969822: 20 mg LY2969822 administered once, PO.
- Cohort 1 - 40 mg LY2969822: 40 mg LY2969822 administered once, PO.
- Cohort 2 - 6 mg LY2969822: 6 mg LY2969822 administered once, PO.
- Cohort 2 - 60 mg LY2969822: 60 mg LY2969822 administered once, PO.
- Cohorts 3-7 - Placebo: Placebo administered QD or BID, PO, for 14 days.
Arm/Group | Cohort 1 - Placebo | Cohort 1 - 2 mg LY2969822 | Cohort 1 - 20 mg LY2969822 | Cohort 1 - 40 mg LY2969822 | Cohort 2 - Placebo | Cohort 2 - 6 mg LY2969822 | Cohort 2 - 60 mg LY2969822 | Cohort 2 - 20 mg LY2969822 | Cohorts 3-7 - Placebo | Cohort 3 - 20 mg LY2969822 QD | Cohort 4 - 40 mg LY2969822 QD Titrated | Cohort 5 - 80 mg LY2969822 QD Titrated | Cohort 6 - 80 mg LY2969822 BID Titrated | Cohort 7 - 40 mg LY2969822 BID Rapidly Titrated | Cohort 8 - Placebo BID | Cohort 8A - 40 mg LY2969822 BID Titrated | Cohort 8B - 20 mg LY2969822 BID Titrated
Number analyzed (Participants) | 9 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 15 | 9 | 9 | 9 | 9 | 9 | 10 | 4 | 7
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Plasma Cmax) of Prodrug LY2969822 and Active Metabolite LSN2934747
Description: Pharmacokinetics (PK): Maximum Plasma Concentration (Plasma Cmax) of Prodrug LY2969822 and Active Metabolite LSN2934747
Time Frame: All Cohorts: Day 1 - 0 Hours (H), 0.5 H, 1 H, 2 H, 3 H, 4 H, 6 H, 9 H, 12 H, 16 H; Cohort 3: Day 10 - 0 H, 0.5 H, 1 H, 2 H, 3 H, 4 H, 6 H, 9 H, 12 H, 16 H; Cohorts 3 - 8: Day 14 - 0 H, 0.5 H,1 H, 2 H, 3 H, 4 H, 6 H, 9 H, 12 H, 16 H
Population: All participants who received at least one dose of LY2969822 and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Groups:
- Cohort 1 - 2 mg LY2969822: 2 mg LY2969822 administered once, PO.
- Cohort 3 - 20 mg LY2969822 QD Day 1 (Fasted); Cohort 3 - 20 mg LY2969822 QD Day 14 (Fasted); Cohort 3 - 20 mg LY2969822 QD Day 10 (Fed): 20 mg LY2969822 administered QD, PO, for 14 days.
- Cohort 4 - 6 mg LY2969822 QD Day 1; Cohort 4 - 40 mg LY2969822 QD Day 14: 6 mg up to 40 mg LY2969822 administered QD, PO, for 14 days. Titration: 6 mg QD for 3 days, 20 mg QD for 2 days, and 40 mg QD for 9 days.
- Cohort 5 - 6 mg LY2969822 QD Day 1; Cohort 5 - 80 mg LY2969822 QD Day 14: 6 mg up to 80 mg LY2969822 administered QD, PO, for 14 days. Titration: 6 mg QD for 2 days, 20 mg QD for 2 days, 40 mg QD for 2 days and 80 mg QD for 8 days.
- Cohort 6 - 6 mg LY2969822 BID Day 1; Cohort 6 - 80 mg LY2969822 BID Day 14: 6 mg up to 80 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, 40 mg BID for 2 days, and 80 mg BID for 6 days.
- Cohort 7 - 10 mg LY2969822 BID Day 1; Cohort 7 - 40 mg LY2969822 BID Day 14: 10 mg up to 40 mg LY2969822 administered QD, PO, for 14 days. Titration: 10 mg BID for 1 day, 20 mg BID for 1 day, and 40 mg BID for 12 days.
- Cohort 8A - 6 mg LY2969822 BID Day 1; Cohort 8A - 40 mg BID LY2969822 Day 14: 6 mg up to 40 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, and 40 mg BID for 8 days.
- Cohort 8B - 6 mg LY2969822 BID Day 1; Cohort 8B - 20 mg BID LY2969822 Day 14: 6 mg up to 20 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 10 days.
Arm/Group | Cohort 1 - 2 mg LY2969822 | Cohort 1 - 20 mg LY2969822 | Cohort 1 - 40 mg LY2969822 | Cohort 2 - 6 mg LY2969822 | Cohort 2 - 60 mg LY2969822 | Cohort 2 - 20 mg LY2969822 | Cohort 3 - 20 mg LY2969822 QD Day 1 (Fasted) | Cohort 3 - 20 mg LY2969822 QD Day 14 (Fasted) | Cohort 3 - 20 mg LY2969822 QD Day 10 (Fed) | Cohort 4 - 6 mg LY2969822 QD Day 1 | Cohort 4 - 40 mg LY2969822 QD Day 14 | Cohort 5 - 6 mg LY2969822 QD Day 1 | Cohort 5 - 80 mg LY2969822 QD Day 14 | Cohort 6 - 6 mg LY2969822 BID Day 1 | Cohort 6 - 80 mg LY2969822 BID Day 14 | Cohort 7 - 10 mg LY2969822 BID Day 1 | Cohort 7 - 40 mg LY2969822 BID Day 14 | Cohort 8A - 6 mg LY2969822 BID Day 1 | Cohort 8A - 40 mg BID LY2969822 Day 14 | Cohort 8B - 6 mg LY2969822 BID Day 1 | Cohort 8B - 20 mg BID LY2969822 Day 14
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 9 | 8 | 9 | 9 | 8 | 9 | 8 | 9 | 8 | 9 | 5 | 4 | 1 | 7 | 6
nanomoles per liter (nmol/L)
  LY2969822 | 19.9 (28) | 209 (20) | 346 (21) | 63.3 (33) | 646 (31) | 197 (22) | 192 (47) | 216 (33) | 341 (33) | 51.3 (67) | 340 (35) | 60.2 (28) | 771 (51) | 49.8 (34) | 788 (30) | 85.9 (43) | 539 (35) | 61.3 (59) | NA (NA) — n=1. Individual value is 467.45 nmol/L. | 44.9 (35) | 216 (32)
  LSN2934747 | 108 (21) | 978 (10) | 1700 (19) | 289 (43) | 2850 (18) | 840 (20) | 847 (30) | 1200 (18) | 1520 (14) | 232 (35) | 1600 (20) | 332 (31) | 4190 (28) | 303 (35) | 4130 (14) | 461 (50) | 2390 (17) | 381 (21) | NA (NA) — n=1. Individual value is 2777.08 nmol/L. | 263 (29) | 1150 (14)

3. Secondary Outcome: PK: Maximum Cerebrospinal Fluid Concentrations (CSF Cmax) of Prodrug LY2969822 and Active Metabolite LSN2934747
Description: PK: Maximum Cerebrospinal Fluid Concentrations (CSF Cmax) of Prodrug LY2969822 and Active Metabolite LSN2934747
Time Frame: Cohort 8: Day 14 - 0 H, 0.5 H,1 H, 2 H, 3 H, 4 H, 6 H, 9 H, 12 H, 16 H
Population: CSF samples were only collected in Cohort 8. All participants in Cohort 8 who received at least one dose of LY2969822 and had evaluable CSF values on Day 14.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Cohort 8A - 40 mg BID LY2969822 Day 14 | Cohort 8B - 20 mg BID LY2969822 Day 14
Number analyzed (Participants) | 1 | 6
nmol/L
  LY2969822 | NA (NA) — n=1. Individual value is 9.86 nmol/L. | 8.42 (106)
  LSN2934747 | NA (NA) — n=1. Individual value is 149 nmol/L. | 93.0 (59)

4. Secondary Outcome: PK: Area Under the Drug Plasma Concentration Time Curve (Plasma AUC) of Prodrug LY2969822 and Active Metabolite LSN2934747
Description: For Cohorts 1-2, AUC is extrapolated from time zero to infinity (AUC[0-inf]). For Cohorts 3 - 8, AUC is reported during one dosing interval (AUC[tau]). AUC(tau) is 24 hours for Cohorts 3 - 5 and 12 hours for Cohorts 6 - 8.
Time Frame: as for outcome 2
Population: All participants who received at least one dose of LY2969822 and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles x hours per liter (nmol∙h/L)
Groups:
- Cohort 8B - 6 mg BID Day 1; Cohort 8B - 20 mg BID Day 14: 6 mg up to 40 mg LY2969822 administered BID, PO, for 14 days. Titration: 6 mg BID for 2 days, 10 mg BID for 2 days, 20 mg BID for 2 days, and 40 mg BID for 8 days.
Arm/Group | Cohort 1 - 2 mg LY2969822 | Cohort 1 - 20 mg LY2969822 | Cohort 1 - 40 mg LY2969822 | Cohort 2 - 6 mg LY2969822 | Cohort 2 - 60 mg LY2969822 | Cohort 2 - 20 mg LY2969822 | Cohort 3 - 20 mg LY2969822 QD Day 1 (Fasted) | Cohort 3 - 20 mg LY2969822 QD Day 14 (Fasted) | Cohort 3 - 20 mg LY2969822 QD Day 10 (Fed) | Cohort 4 - 6 mg LY2969822 QD Day 1 | Cohort 4 - 40 mg LY2969822 QD Day 14 | Cohort 5 - 6 mg LY2969822 QD Day 1 | Cohort 5 - 80 mg LY2969822 QD Day 14 | Cohort 6 - 6 mg LY2969822 BID Day 1 | Cohort 6 - 80 mg LY2969822 BID Day 14 | Cohort 7 - 10 mg LY2969822 BID Day 1 | Cohort 7 - 40 mg LY2969822 BID Day 14 | Cohort 8A - 6 mg LY2969822 BID Day 1 | Cohort 8A - 40 mg BID LY2969822 Day 14 | Cohort 8B - 6 mg BID Day 1 | Cohort 8B - 20 mg BID Day 14
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 9 | 8 | 9 | 9 | 8 | 9 | 8 | 9 | 8 | 9 | 5 | 4 | 1 | 7 | 6
nanomoles x hours per liter (nmol∙h/L)
  LY2969822 | 88.5 (22) | 843 (19) | 1730 (12) | 273 (36) | 3700 (26) | 1110 (38) | 759 (50) | 896 (27) | 1160 (25) | 231 (51) | 1400 (42) | 244 (36) | 3430 (55) | 203 (42) | 2810 (35) | 363 (46) | 1820 (40) | 306 (65) | NA (NA) — n=1. Individual value is 1840 nmol∙h/L. | 207 (44) | 778 (34)
  LSN2934747 | 805 (18) | 7030 (12) | 13500 (25) | 2090 (39) | 23600 (17) | 6970 (22) | 5830 (36) | 8220 (15) | 8660 (12) | 1710 (28) | 10600 (28) | 2100 (26) | 29000 (30) | 1810 (30) | 25300 (18) | 3010 (49) | 14400 (19) | 2670 (20) | NA (NA) — n=1. Individual value is 15800 nmol∙h/L. | 1790 (20) | 6920 (18)

5. Secondary Outcome: PK: CSF AUC(Tau) of Prodrug LY2969822 and Active Metabolite LSN2934747
Description: AUC(tau) is 12 hours.
Time Frame: Cohort 8: Day 14 - 0 H, 0.5 H,1 H, 2 H, 3 H, 4 H, 6 H, 9 H, 12 H, 16 H
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol∙h/L
Arm/Group | Cohort 8A - 40 mg BID LY2969822 Day 14 | Cohort 8B - 20 mg BID LY2969822 Day 14
Number analyzed (Participants) | 1 | 6
nmol∙h/L
  LY2969822 | NA (NA) — n=1. Individual value is 1840 nmol∙h/L. | 75.1 (85)
  LSN2934747 | NA (NA) — n=1. Individual value is 15800 nmol∙h/L. | 831 (61)

ADVERSE EVENTS:
Groups:
- Part A: Placebo: Placebo administered once, PO.
- Part A: 2 mg LY2969822: 2 mg LY2969822 administered once, PO.
- Part A: 6 mg LY2969822: 6 mg LY2969822 administered once, PO.
- Part A: 20 mg LY2969822: 20 mg LY2969822 administered once, PO.
- Part A: 40 mg LY2969822: 40 mg LY2969822 administered once, PO.
- Part A: 60 mg LY2969822: 60 mg LY2969822 administered once, PO.
- Part B: Placebo: Placebo administered QD, PO, for 14 days.
- Part B: Placebo BID; Part C: Placebo BID: Placebo administered BID, PO, for 14 days.
- Part B: 6 mg LY2969822: 6 mg LY2969822 administered QD, PO, for 2 - 3 days
- Part B: 6 mg LY2969822 BID; Part C: 6 mg LY2969822 BID: 6 mg LY2969822 administered BID, PO, for 2 days.
- Part B: 10 mg LY2969822 BID: 10 mg LY2969822 administered BID, PO, for 1-2 days.
- Part B: 20 mg LY2969822: 20 mg LY2969822 administered QD, PO, for up to 14 days.
- Part B: 20 mg LY2969822 BID: 20 mg LY2969822 administered BID, PO, for 1-2 days.
- Part B: 40 mg LY2969822: 40 mg LY2969822 administered QD, PO, for up to 9 days.
- Part B: 40 mg LY2969822 BID: 40 mg LY2969822 administered BID, PO, for up to 12 days.
- Part B: 80 mg LY2969822: 80 mg LY2969822 administered QD, PO, for 8 days.
- Part B: 80 mg LY2969822 BID: 80 mg LY2969822 administered BID, PO, for 6 days.
- Part C: 10 mg LY2969822 BID: 10 mg LY2969822 administered BID, PO, for 2 days.
- Part C: 20 mg LY2969822 BID: 20 mg LY2969822 administered BID, PO, for up to 10 days.
- Part C: 40 mg LY2969822 BID: 40 mg LY2969822 administered BID, PO, for up to 8 days.
Arm/Group | Part A: Placebo | Part A: 2 mg LY2969822 | Part A: 6 mg LY2969822 | Part A: 20 mg LY2969822 | Part A: 40 mg LY2969822 | Part A: 60 mg LY2969822 | Part B: Placebo | Part B: Placebo BID | Part B: 6 mg LY2969822 | Part B: 6 mg LY2969822 BID | Part B: 10 mg LY2969822 BID | Part B: 20 mg LY2969822 | Part B: 20 mg LY2969822 BID | Part B: 40 mg LY2969822 | Part B: 40 mg LY2969822 BID | Part B: 80 mg LY2969822 | Part B: 80 mg LY2969822 BID | Part C: Placebo BID | Part C: 6 mg LY2969822 BID | Part C: 10 mg LY2969822 BID | Part C: 20 mg LY2969822 BID | Part C: 40 mg LY2969822 BID
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/12 | 0/5 | 0/6 | 0/9 | 0/6 | 0/18 | 0/9 | 0/18 | 0/27 | 0/17 | 0/18 | 0/16 | 0/9 | 0/8 | 0/10 | 0/11 | 0/11 | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 5/18 | 3/6 | 4/6 | 8/12 | 4/5 | 6/6 | 8/9 | 5/6 | 12/18 | 8/9 | 17/18 | 21/27 | 16/17 | 16/18 | 15/16 | 8/9 | 8/8 | 10/10 | 10/11 | 10/11 | 11/11 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=18) | Part A: 2 mg LY2969822 (N=6) | Part A: 6 mg LY2969822 (N=6) | Part A: 20 mg LY2969822 (N=12) | Part A: 40 mg LY2969822 (N=5) | Part A: 60 mg LY2969822 (N=6) | Part B: Placebo (N=9) | Part B: Placebo BID (N=6) | Part B: 6 mg LY2969822 (N=18) | Part B: 6 mg LY2969822 BID (N=9) | Part B: 10 mg LY2969822 BID (N=18) | Part B: 20 mg LY2969822 (N=27) | Part B: 20 mg LY2969822 BID (N=17) | Part B: 40 mg LY2969822 (N=18) | Part B: 40 mg LY2969822 BID (N=16) | Part B: 80 mg LY2969822 (N=9) | Part B: 80 mg LY2969822 BID (N=8) | Part C: Placebo BID (N=10) | Part C: 6 mg LY2969822 BID (N=11) | Part C: 10 mg LY2969822 BID (N=11) | Part C: 20 mg LY2969822 BID (N=11) | Part C: 40 mg LY2969822 BID (N=4)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (36) | 2 (2) | 4 (5) | 6 (12) | 2 (2) | 7 (9) | 2 (2) | 6 (10) | 2 (2) | 5 (16) | 7 (23) | 5 (7) | 10 (13) | 8 (13) | 4 (8)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 1 (3) | 1 (2) | 9 (16) | 4 (4) | 7 (8) | 9 (15) | 3 (5) | 6 (9) | 4 (5) | 3 (3) | 0 (0) | 2 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 6 (27) | 0 (0) | 0 (0) | 4 (12) | 2 (3) | 4 (20) | 8 (33) | 2 (5) | 5 (25) | 3 (12) | 3 (8) | 1 (4) | 2 (6) | 3 (5) | 0 (0) | 1 (3) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (11) | 3 (7) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 4 (8) | 6 (9) | 1 (1) | 2 (2) | 3 (6) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (4)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 2 (2) | 1 (1) | 2 (3) | 4 (5) | 3 (4) | 6 (6) | 10 (20) | 5 (7) | 4 (6) | 8 (12) | 3 (5) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (11) | 1 (4) | 2 (3) | 1 (1) | 1 (1) | 7 (13) | 1 (2) | 5 (6) | 6 (11) | 2 (3) | 3 (3) | 5 (7) | 2 (2) | 0 (0) | 4 (7) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes